CLINICAL TRIAL: NCT01934023
Title: Effects of Varenicline on Cortical Neuroplasticity and Working Memory in Patients With Schizophrenia and Healthy Controls
Brief Title: Effects of Varenicline on Plasticity in Schizophrenia
Acronym: VAR-PAS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre for Addiction and Mental Health (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Principal Investigator, Tony George, Chief, Schizophrenia Division, Centre for Addiction and Mental Health
Allocation: Randomized | Model: Crossover | Masking: Double
Other Study IDs: 214-2012; Wi172662 (Other Grant/Funding Number: Pfizer)
Record Dates: First submitted 2013-08-27; First posted 2013-09-04 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Schizophrenia
Keywords: plasticity, schizophrenia, varenicline, non smokers,
MeSH Terms: conditions — Schizophrenia | interventions — Varenicline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Varenicline (Active Comparator): FDA approved smoking cessation medication
  Interventions: Drug: Varenicline
- Placebo Sugar Pill (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Varenicline — Champix (Varenicline) is an approved smoking cessation medication
  Other Names: Champix
  Arms: Varenicline
Drug: Placebo
  Arms: Placebo Sugar Pill

SUMMARY:
This laboratory pilot study will explore the effects of varenicline tartrate on long-term potentiation (LTP)-like mechanisms of (1) the motor cortex and (2) the dorsolateral prefrontal cortex (DLPFC) and working memory in non-smoking patients with schizophrenia and healthy controls using a Paired Associative Stimulation (PAS) method. The present study will use this novel PAS method to evaluate the effects of five doses of varenicline (Champix) 0.5 mg BID treatment on neuroplasticity changes and working memory in 28 non-smokers with schizophrenia and 28 non-smoking controls in a placebo-controlled, double-blinded, cross-over design. The hypothesis is that varenicline will increase LTP-like facilitation of the DLPFC as compared with placebo in patients with schizophrenia, with less or a null effect in healthy controls. Likewise, it is hypothesized that varenicline will specifically improve working memory in patients with schizophrenia as compared with placebo and healthy controls. We Hypothesize that: 1.Patients with Schizophrenia(SCZ) will have reduced cortical LTP and impaired working memory compared to healthy controls 2. Sub-chronic varenicline challenge will attenuate the cortical LTP and working memory deficit in patients with SCZ. 3.Reversal of the cortical LTP deficit by varenicline in patients with SCZ will be associated with improvement in working memory.

DETAILED DESCRIPTION:
The experimental laboratory study will be designed as a randomized, double-blinded, placebo-controlled acute treatment trial. Paired Associative Stimulation (PAS)-induced cortical evoked activity and Working Memory (WM) will be assessed in healthy non-smokers and non-smokers with SCZ, after five doses of varenicline tartrate (0.5 mg/dose) and placebo treatment. PAS will be induced by pairing transcranial magnetic stimulation with peripheral nerve stimulation, 25 msec apart (hence PAS-25). In part 1, motor cortex plasticity will be assessed as changes in motor evoked potential comparing pre to post PAS up tp 120 min after PAS. In part 2, DLPFC evoked cortical activity will be assessed using EEG comparing pre to post PAS. Effects of varenicline and PAS-25 on WM will evaluated using a computerized N-back task, assessed directly before the PAS testing. The whole experimental session will be repeated for each participant twice: once with varenicline tartrate treatment and once with placebo treatment, two weeks apart.

ELIGIBILITY:
Inclusion Criteria (Healthy subjects and Scz):

* Non-smoker or past smoker, abstinent for at least the last 1 year
* Females with potential childbearing must have a negative serum pregnancy test at inclusion.
* Ability and willingness to speak English
* Willingness to provide informed consent
* Adequate hearing and visual capacity, or corrected by visual/ hearing aid, right handedness.

INCLUSION Criteria (Scz Only):

* Diagnosis of schizophrenia
* Stable psychotropic drug treatment for at least the past 4 weeks
* Clinically stable for the past 3 months.

Exclusion Criteria (healthy subjects and SCZ):

* Current smoker or abstinent smoker for less than 1 year
* Current history of drug abuse disorder or current elicit drug use
* Current or past history of neurological disorder
* Current or past history of seizures
* Any metal implants
* Mini Mental Status Examination score of less than 20
* Diagnosis of bipolar disorder or current Major depression episode
* Electroconvulsive Therapy (ECT) within 6 months
* Varenicline hypersensitivity.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2013-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Change of Paired Associative Stimulation (PAS) induced plasticity from baseline | Day 3 of weeks 1 and 2

SECONDARY OUTCOMES:
Change of Working memory performance from baseline | Day 3 of weeks 1 and 2

CONTACTS AND LOCATIONS:
Overall Officials: Tony P George, M.D, Principal Investigator — Centre for Addiction Mental Health
Locations (1):
- Centre for Addiction and Mental Health, Toronto, Ontario, Canada

REFERENCES:
- See also: Centre for Addiction and Mental Health Research — http://www.camh.net/research